CLINICAL TRIAL: NCT02476890
Title: A Study to Assess the Effect of MK-7264 (AF-219) on Cough Reflex Sensitivity in Both Healthy and Chronic Cough Subjects
Brief Title: Effect of Gefapixant (MK-7264/AF-219) on Cough Reflex Sensitivity in Healthy and Chronic Cough Participants (MK-7264-014)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Afferent Pharmaceuticals, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 7264-014; MK-7264-014 (Other: Merck Protocol Number); AF-219-014 (Other: Afferent Protocol Number); 2015-002034-47 (EudraCT Number); NCT03407014 (obsolete NCT alias)
Record Dates: First submitted 2015-06-15; First posted 2015-06-22 (Estimated); Results first posted 2018-02-15 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Refractory Chronic Cough
MeSH Terms: conditions — Chronic Cough | interventions — Gefapixant

STUDY DESIGN:
Intervention Model Description: Chronic cough and healthy participants were randomly assigned to receive gefapixant and placebo in one of two treatment sequences: Sequence A (placebo in treatment period 1, then gefapixant in treatment period 2) or Sequence B (gefapixant in treatment period 1, then placebo in treatment period 2). There was at least a 48-hour washout between the treatment periods. Daytime cough monitoring was performed in chronic cough participants only.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Placebo then gefapixant 100 mg/Healthy (Sequence A) (Experimental): Healthy participants in Sequence A received a single dose of placebo in treatment Period 1 then a single dose of gefapixant 100 mg in treatment Period 2. There was a minimum 48-hr washout between Periods 1 & 2.
  Interventions: Drug: Gefapixant 100 mg; Drug: Placebo
- Gefapixant 100 mg then placebo/Healthy (Sequence B) (Experimental): Healthy participants in Sequence B received a single dose of gefapixant 100 mg in treatment Period 1 then a single dose of placebo in treatment Period 2. There was a minimum 48-hr washout between Periods 1 & 2.
  Interventions: Drug: Gefapixant 100 mg; Drug: Placebo
- Placebo then gefapixant 100 mg/Chronic Cough (Sequence A) (Experimental): Chronic Cough participants in Sequence A received a single dose of placebo in treatment Period 1 then a single dose of gefapixant 100 mg in treatment Period 2. There was a minimum 48-hr washout between Periods 1 & 2.
  Interventions: Drug: Gefapixant 100 mg; Drug: Placebo
- Gefapixant 100 mg then placebo/Chronic Cough (Sequence B) (Experimental): Chronic Cough participants in Sequence B received a single dose of gefapixant 100 mg in treatment Period 1 then a single dose of placebo in treatment Period 2. There was a minimum 48-hr washout between Periods 1 & 2.
  Interventions: Drug: Gefapixant 100 mg; Drug: Placebo

INTERVENTIONS:
Drug: Gefapixant 100 mg — Gefapixant 100 mg (2 x 50 mg tablets), administered orally as a single dose in treatment Period 1 or treatment Period 2
  Other Names: MK-7264; AF-219
Drug: Placebo — Placebo (two tablets matching gefapixant 50 mg), administered orally as a single dose in treatment Period 1 or treatment Period 2

SUMMARY:
The primary objective of this study was to assess the effect of a single dose of gefapixant 100 mg on cough reflex sensitivity to various challenge agents (capsaicin, citric acid, adenosine triphosphate [ATP], and distilled water) in healthy and chronic cough participants.

DETAILED DESCRIPTION:
The study had a Screening period to determine participant inclusion, two Baseline Visits, and two treatment periods with a minimum 48-hour washout between the treatment periods. At Baseline and during each treatment period, cough sensitivity was measured by standard clinical methodology incorporating four cough challenges. Daytime cough monitoring was performed at Baseline and during each of the two treatment periods (chronic cough participants only).

ELIGIBILITY:
Inclusion Criteria:

* Have provided written informed voluntary consent;
* Be able to speak, read, and understand English;
* Be males or females, of any race, between 18 and 80 years of age, inclusive;
* Have a body mass index (BMI) >= 18 and < 35 kg/m^2;
* Be in good general health with no clinically relevant abnormalities based on the medical history, physical examination, clinical laboratory evaluations (hematology, clinical chemistry, and urinalysis), and 12 lead electrocardiogram;
* Be non-smokers for at least 5 years;
* If a female of child-bearing potential (I. e., have not undergone a hysterectomy or bilateral oophorectomy) or not post-menopausal (defined as no menses for at least 12 months), agree to use 2 forms of acceptable birth control; or if a male, they and/or their partner of child-bearing potential agree to use 2 forms of acceptable birth control;
* Be able to communicate effectively with the Investigator and other study center personnel and agree to comply with the study procedures and restrictions.
* Subjects with chronic cough must have treatment-refractory chronic cough for at least one year, with no objective evidence of an underlying trigger (e. g., asthma)

Exclusion Criteria:

* History of upper respiratory tract infection or recent significant change in pulmonary status within 4 weeks of the Baseline Visit (Day 0);
* Have acute worsening of asthma;
* Do not cough during the ATP or Capsaicin or Citric acid challenge at Screening or only cough twice at the two highest concentrations of the test solution;
* History of concurrent malignancy or recurrence of malignancy within 2 years prior to Screening (not including subjects with <3 excised basal cell carcinomas);
* History of a diagnosis of drug or alcohol dependency or abuse within approximately the last 3 years;
* Clinically significant abnormal electrocardiogram (ECG) at Screening;
* Significantly abnormal laboratory tests at Screening;
* Pregnant or breastfeeding;
* Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the Investigator or Sponsor, would make the subject inappropriate for entry into this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2016-10-20 (Actual); Study Completion 2016-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Morice AH, Kitt MM, Ford AP, Tershakovec AM, Wu WC, Brindle K, Thompson R, Thackray-Nocera S, Wright C. The effect of gefapixant, a P2X3 antagonist, on cough reflex sensitivity: a randomised placebo-controlled study. Eur Respir J. 2019 Jul 4;54(1):1900439. doi: 10.1183/13993003.00439-2019. Print 2019 Jul. PMID 31023843

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A 6-day Screening period (Day -6 to Day -1) ensured that each participant met all the specified eligibility criteria. In addition, cough reflex sensitivity was measured at Screening by standard clinical methodology using cough challenge in response to four agents (capsaicin, citric acid, adenosine triphosphate (ATP), and distilled water).
Groups:
- Placebo Then Gefapixant 100 mg/Healthy (Sequence A): Healthy participants in Sequence A received a single dose of placebo in treatment Period 1 then a single dose of gefapixant 100 mg in treatment Period 2. There was a washout period of at least 48 hours between Period 1 and Period 2.
- Gefapixant 100 mg Then Placebo/Healthy (Sequence B): Healthy participants in Sequence B received a single dose of gefapixant 100 mg in treatment Period 1 then a single dose of placebo in treatment Period 2. There was a washout period of at least 48 hours between Period 1 and Period 2.
- Placebo Then Gefapixant 100 mg/Chronic Cough (Sequence A): Chronic Cough participants in Sequence A received a single dose of placebo in treatment Period 1 then a single dose of gefapixant 100 mg in treatment Period 2. There was a washout period of at least 48 hours between Period 1 and Period 2.
- Gefapixant 100 mg Then Placebo/Chronic Cough (Sequence B): Chronic Cough participants in Sequence B received a single dose of gefapixant 100 mg in treatment Period 1 then a single dose of placebo in treatment Period 2. There was a washout period of at least 48 hours between Period 1 and Period 2.
Period: Overall Study
Arm/Group | Placebo Then Gefapixant 100 mg/Healthy (Sequence A) | Gefapixant 100 mg Then Placebo/Healthy (Sequence B) | Placebo Then Gefapixant 100 mg/Chronic Cough (Sequence A) | Gefapixant 100 mg Then Placebo/Chronic Cough (Sequence B)
Started | 6 (Crossover study) | 6 (Crossover study) | 12 (Crossover study) | 12 (Crossover study)
Washout | 6 | 6 | 12 | 12
Completed | 6 | 6 | 12 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Then Gefapixant 100 mg/Healthy (Sequence A): Healthy participants in Sequence A were randomized to receive placebo in treatment Period 1, then gefapixant 100 mg in treatment Period 2.
- Gefapixant 100 mg Then Placebo/Healthy (Sequence B): Healthy participants in Sequence B were randomized to receive gefapixant 100 mg in treatment Period 1, then placebo in treatment Period 2.
- Placebo Then Gefapixant 100 mg/Chronic Cough (Sequence A): Chronic Cough Participants in Sequence A were randomized to receive placebo in treatment Period 1, then gefapixant 100 mg in treatment Period 2.
- Gefapixant 100 mg Then Placebo/Chronic Cough (Sequence B): Chronic Cough participants in Sequence B were randomized to receive gefapixant 100 mg in treatment Period 1, then placebo in treatment Period 2.
- Total: Total of all reporting groups
Arm/Group | Placebo Then Gefapixant 100 mg/Healthy (Sequence A) | Gefapixant 100 mg Then Placebo/Healthy (Sequence B) | Placebo Then Gefapixant 100 mg/Chronic Cough (Sequence A) | Gefapixant 100 mg Then Placebo/Chronic Cough (Sequence B) | Total
Number analyzed (Participants) | 6 | 6 | 12 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (10.79) | 35.7 (6.09) | 61.6 (9.15) | 60.6 (8.58) | 53.3 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11 | 10 | 32
  Male | 0 | 1 | 1 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Cough Reflex Sensitivity to Capsaicin in Participants Who Received Gefapixant 100 mg and Placebo (Period 1 & Period 2 Combined)
Description: The concentration of capsaicin inducing at least 2 coughs (C2) and at least 5 coughs (C5) was assessed at 1, 3, and 5 hours post-dose in healthy and chronic cough participants. The concentrations of capsaicin for cough challenge were 0.3 micromoles (µM), 1 µM, 3 µM, 10 µM, 30 µM, 100 µM, 300 µM, and 1000 µM. The Measure Type is least-squares mean in natural log scale. The challenge agent was prepared by dilution of capsaicin with saline, and was administered by inhalation. A mixed effects model used natural log-transformed values for the lowest concentrations of inhaled solution required to evoke at least 2 (C2) or at least 5 (C5) coughs to estimate the average of C2 or C5 across 3 time points for each treatment group, and to compare treatment difference relative to placebo. When applying the mixed model repeated measure analysis, if there is a missing value for concentration, it was imputed as 1.5 times the maximum concentration (=150%).
Time Frame: Average of 1, 3, and 5 hours post-dose
Population: The analyzed population was all treated participants who had at least 1 post-dose primary endpoint assessment of cough reflex sensitivity in response to capsaicin challenge.
Measure: Least Squares Mean (95% Confidence Interval); unit: natural log (µM)
Groups:
- Gefapixant 100 mg/Healthy: Healthy participants received a single dose of gefapixant 100 mg in Period 1 or Period 2, with crossover to or from placebo following a minimum 48-hour washout.
- Placebo/Healthy: Healthy participants received a single dose of placebo in Period 1 or Period 2, with crossover to or from gefapixant 100 mg following a minimum 48-hour washout.
- Gefapixant 100 mg/Chronic Cough: Chronic Cough participants received a single dose of gefapixant 100 mg in Period 1 or Period 2, with crossover to or from placebo following a minimum 48-hour washout.
- Placebo/Chronic Cough: Chronic Cough participants received a single dose of placebo in Period 1 or Period 2, with crossover to or from gefapixant 100 mg following a minimum 48-hour washout.
Arm/Group | Gefapixant 100 mg/Healthy | Placebo/Healthy | Gefapixant 100 mg/Chronic Cough | Placebo/Chronic Cough
Number analyzed (Participants) | 12 | 12 | 24 | 24
natural log (µM)
  C2 Response to Capsaicin (Periods 1 & 2) | 3.05 [2.6 to 3.5] | 3.04 [2.6 to 3.5] | 1.72 [1.3 to 2.1] | 1.41 [1.0 to 1.8]
  C5 Response to Capsaicin (Periods 1 & 2) | 4.46 [3.9 to 5.0] | 4.68 [4.1 to 5.3] | 2.31 [1.9 to 2.8] | 2.05 [1.6 to 2.5]
Statistical Analysis 1: Comparison: Gefapixant 100 mg/Healthy vs Placebo/Healthy; C2 Response/Healthy; Test type: Other; p = 0.9666, Mixed Models Analysis; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.6 to 0.7]
Statistical Analysis 2: Comparison: Gefapixant 100 mg/Healthy vs Placebo/Healthy; C5 Response/Healthy; Test type: Other; p = 0.5993, Mixed Models Analysis; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-1.1 to 0.6]
Statistical Analysis 3: Comparison: Gefapixant 100 mg/Chronic Cough vs Placebo/Chronic Cough; C2 Response/Chronic Cough; Test type: Other; p = 0.2823, Mixed Models Analysis; Mean Difference (Final Values) = 0.32, 95% CI 2-sided [-0.3 to 0.9]
Statistical Analysis 4: Comparison: Gefapixant 100 mg/Chronic Cough vs Placebo/Chronic Cough; C5 Response/Chronic Cough; Test type: Other; p = 0.4287, Mixed Models Analysis; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [-0.4 to 0.9]

2. Primary Outcome: Cough Reflex Sensitivity to Citric Acid in Participants Who Received Gefapixant 100 mg and Placebo (Period 1 & Period 2 Combined)
Description: The concentration of citric acid inducing at least 2 coughs (C2) and at least 5 coughs (C5) was assessed at 1, 3, and 5 hours post-dose in healthy and chronic cough participants. The concentrations of citric acid for cough challenge were 1 millimoles (mM), 3 mM, 10 mM, 30 mM, 100 mM, 300 mM, 1 M, and 3 M. The Measure Type is least-squares mean in natural log scale. The challenge agent was prepared by dilution of citric acid with saline, and was administered by inhalation. A mixed effects model used natural log-transformed values for the lowest concentrations of inhaled solution required to evoke at least 2 (C2) or at least 5 (C5) coughs to estimate the average of C2 or C5 across 3 time points for each treatment group, and to compare treatment difference relative to placebo. When applying the mixed model repeated measure analysis, if there is a missing value for concentration, it was imputed as 1.5 times the maximum concentration (=150%).
Time Frame: Average of 1, 3, and 5 hours post-dose
Population: The analyzed population was all treated participants who had at least 1 post-dose primary endpoint assessment of cough reflex sensitivity in response to citric acid challenge.
Measure: Least Squares Mean (95% Confidence Interval); unit: natural log (mM)
Arm/Group | Gefapixant 100 mg/Healthy | Placebo/Healthy | Gefapixant 100 mg/Chronic Cough | Placebo/Chronic Cough
Number analyzed (Participants) | 12 | 12 | 24 | 24
natural log (mM)
  C2 Response to Citric Acid (Periods 1 & 2) | 6.16 [5.6 to 6.8] | 5.61 [5.0 to 6.2] | 4.07 [3.6 to 4.6] | 3.84 [3.3 to 4.3]
  C5 Response to Citric Acid (Periods 1 & 2) | 7.12 [6.4 to 7.8] | 6.82 [6.1 to 7.6] | 4.74 [4.2 to 5.2] | 4.46 [4.0 to 5.0]
Statistical Analysis 1: Comparison: Gefapixant 100 mg/Healthy vs Placebo/Healthy; C2 Response/Healthy; Test type: Other; p = 0.1771, Mixed Models Analysis; Mean Difference (Final Values) = 0.56, 95% CI 2-sided [-0.3 to 1.4]
Statistical Analysis 2: Comparison: Gefapixant 100 mg/Healthy vs Placebo/Healthy; C5 Response/Healthy; Test type: Other; p = 0.5473, Mixed Models Analysis; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.7 to 1.3]
Statistical Analysis 3: Comparison: Gefapixant 100 mg/Chronic Cough vs Placebo/Chronic Cough; C2 Response/Chronic Cough; Test type: Other; p = 0.5169, Mixed Models Analysis; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-0.5 to 1.0]
Statistical Analysis 4: Comparison: Gefapixant 100 mg/Chronic Cough vs Placebo/Chronic Cough; C5 Response/Chronic Cough; Test type: Other; p = 0.4243, Mixed Models Analysis; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-0.4 to 1.0]

3. Primary Outcome: Cough Reflex Sensitivity to ATP in Participants Who Received Gefapixant 100 mg and Placebo (Period 1 & Period 2 Combined)
Description: The concentration of ATP inducing at least 2 coughs (C2) and at least 5 coughs (C5) was assessed at 1, 3, and 5 hours post-dose in healthy and chronic cough participants. The concentrations of ATP for cough challenge were 0.1 mM, 0.3 mM, 1 mM, 3 mM, 10 mM, 30 mM, 100 mM, and 300 mM. The Measure Type is least-squares mean in natural log scale. The challenge agent was prepared by dilution of ATP with saline, and was administered by inhalation. A mixed effects model used natural log-transformed values for the lowest concentrations of inhaled solution required to evoke at least 2 (C2) or at least 5 (C5) coughs to estimate the average of C2 or C5 across 3 time points for each treatment group, and to compare treatment difference relative to placebo. When applying the mixed model repeated measure analysis, if there is a missing value for concentration, it was imputed as 1.5 times the maximum concentration (=150%).
Time Frame: Average of 1, 3, and 5 hours post-dose
Population: The analyzed population was all treated participants who had at least 1 post-dose primary endpoint assessment of cough reflex sensitivity in response to ATP challenge.
Measure: Least Squares Mean (95% Confidence Interval); unit: natural log (mM)
Arm/Group | Gefapixant 100 mg/Healthy | Placebo/Healthy | Gefapixant 100 mg/Chronic Cough | Placebo/Chronic Cough
Number analyzed (Participants) | 12 | 12 | 24 | 24
natural log (mM)
  C2 Response to ATP (Periods 1 & 2) | 4.79 [4.0 to 5.6] | 3.90 [3.1 to 4.7] | 2.90 [2.3 to 3.5] | 1.36 [0.8 to 2.0]
  C5 Response to ATP (Periods 1 & 2) | 5.61 [5.3 to 5.9] | 4.73 [4.3 to 5.1] | 3.52 [2.9 to 4.2] | 2.22 [1.6 to 2.9]
Statistical Analysis 1: Comparison: Gefapixant 100 mg/Healthy vs Placebo/Healthy; C2 Response/Healthy; Test type: Other; p = 0.1125, Mixed Models Analysis; Mean Difference (Final Values) = 0.89, 95% CI 2-sided [-0.2 to 2.0]
Statistical Analysis 2: Comparison: Gefapixant 100 mg/Healthy vs Placebo/Healthy; C5 Response/Healthy; Test type: Other; p = 0.0029, Mixed Models Analysis; Mean Difference (Final Values) = 0.88, 95% CI 2-sided [0.4 to 1.4]
Statistical Analysis 3: Comparison: Gefapixant 100 mg/Chronic Cough vs Placebo/Chronic Cough; C2 Response/Chronic Cough; Test type: Other; p = 0.0006, Mixed Models Analysis; Mean Difference (Final Values) = 1.54, 95% CI 2-sided [0.7 to 2.4]
Statistical Analysis 4: Comparison: Gefapixant 100 mg/Chronic Cough vs Placebo/Chronic Cough; C5 Response/Chronic Cough; Test type: Other; p = 0.0067, Mixed Models Analysis; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [0.4 to 2.2]

4. Primary Outcome: Cough Reflex Sensitivity to Distilled Water in Participants Who Received Gefapixant 100 mg and Placebo (Period 1 & Period 2 Combined)
Description: The concentration of distilled water inducing at least 2 coughs (C2) and at least 5 coughs (C5) was assessed at 1, 3, and 5 hours post-dose in healthy and chronic cough participants. The concentrations of distilled water for cough challenge were 20%, 40%, 60%, 80%, and 100%. The Measure Type is least-squares mean in natural log scale. The number of coughs generated in 1 minute of exposure was recorded. The challenge agent was prepared by dilution of distilled water with saline, and was administered by inhalation. A mixed effects model used natural log-transformed values for the lowest concentrations of inhaled solution required to evoke at least 2 (C2) or at least 5 (C5) coughs to estimate the average of C2 or C5 across 3 time points for each treatment group, and to compare treatment difference relative to placebo. When applying the mixed model repeated measure analysis, if there is a missing value for concentration, it was imputed as 1.5 times the maximum concentration (=150%).
Time Frame: Average of 1, 3, and 5 hours post-dose
Population: The analyzed population was all treated participants who had at least 1 post-dose primary endpoint assessment of cough reflex sensitivity in response to distilled water challenge.
Measure: Least Squares Mean (95% Confidence Interval); unit: natural log (percent concentration [%])
Arm/Group | Gefapixant 100 mg/Healthy | Placebo/Healthy | Gefapixant 100 mg/Chronic Cough | Placebo/Chronic Cough
Number analyzed (Participants) | 12 | 12 | 24 | 24
natural log (percent concentration [%])
  C2 Response to Distilled Water (Periods 1 & 2) | 4.72 [4.6 to 4.8] | 4.34 [4.2 to 4.4] | 4.42 [4.3 to 4.5] | 4.12 [4.0 to 4.2]
  C5 Response to Distilled Water (Periods 1 & 2) | 4.85 [4.6 to 5.1] | 4.61 [4.4 to 4.8] | 4.51 [4.4 to 4.6] | 4.24 [4.1 to 4.4]
Statistical Analysis 1: Comparison: Gefapixant 100 mg/Healthy vs Placebo/Healthy; C2 Response/Healthy; Test type: Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [0.2 to 0.5]
Statistical Analysis 2: Comparison: Gefapixant 100 mg/Healthy; C5 Response/Healthy; Test type: Other; p = 0.1798, Mixed Models Analysis; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-0.1 to 0.6]
Statistical Analysis 3: Comparison: Gefapixant 100 mg/Chronic Cough vs Placebo/Chronic Cough; C2 Response/Chronic Cough; Test type: Other; p = 0.0011, Mixed Models Analysis; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [0.1 to 0.5]
Statistical Analysis 4: Comparison: Gefapixant 100 mg/Chronic Cough vs Placebo/Chronic Cough; C5 Response/Chronic Cough; Test type: Other; p = 0.0023, Mixed Models Analysis; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [0.1 to 0.4]

5. Secondary Outcome: Change From Baseline in Cough Severity Visual Analogue Scale (VAS) After Cough Challenge Testing in Participants Who Received Gefapixant 100 mg and Placebo (Chronic Cough Participants Only)
Description: Chronic cough participants completed a visual analogue scale (VAS) to record cough severity, prior to dosing on the treatment day in each treatment period, and one hour after the final cough challenge on the treatment days. This was a 100mm VAS of cough severity from 'No Cough' (0) up to 'Worst Cough' (100). Participants were instructed to draw a line on the scale to indicate how severe they felt their cough was during the previous 1 hour on the treatment days. A negative change from Baseline was considered to indicate improvement in cough severity.
Time Frame: Baseline and one hour after the final cough challenge on treatment days
Population: The analyzed population was all treated chronic cough participants who had at least 1 post-dose primary endpoint assessment of cough severity.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Gefapixant 100 mg/Chronic Cough | Placebo/Chronic Cough
Number analyzed (Participants) | 24 | 24
Scores on a scale | -26.2 [-36.2 to -16.2] | -8.2 [-18.7 to 2.2]
Statistical Analysis 1: Comparison: Gefapixant 100 mg/Chronic Cough vs Placebo/Chronic Cough; Cough Severity VAS Analysis; Test type: Other; p = 0.0037, Mixed Models Analysis; Mean Difference (Final Values) = -18.0, 95% CI 2-sided [-29.8 to -6.2]

6. Secondary Outcome: Change From Baseline in Urge to Cough VAS After Cough Challenge Testing in Participants Who Received Gefapixant 100 mg and Placebo (Chronic Cough Participants Only)
Description: Chronic cough participants completed a VAS to record the severity of their urge to cough, prior to dosing on the treatment day in each treatment period, and one hour after the final cough challenge on the treatment days. Participants marked the 100mm VAS at the extremes as 'No urge-to-cough' (0) and 'Worst urge-to-cough' (100). Participants were instructed to draw a single vertical line on the scale to indicate how severe their urge to cough was during the previous 1 hour on the treatment days. A negative change from Baseline was considered to indicate improvement in urge to cough.
Time Frame: Baseline and one hour after final cough challenge on treatment days
Population: The analyzed population was all treated chronic cough participants who had at least 1 post-dose primary endpoint assessment of urge to cough.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Gefapixant 100 mg/Chronic Cough | Placebo/Chronic Cough
Number analyzed (Participants) | 24 | 24
Scores on a scale | -29.8 [-38.9 to -20.7] | -11.7 [-20.9 to -2.6]
Statistical Analysis 1: Comparison: Gefapixant 100 mg/Chronic Cough vs Placebo/Chronic Cough; Urge to Cough VAS Analysis; Test type: Other; p = 0.0020, Mixed Models Analysis; Mean Difference (Final Values) = -18.0, 95% CI 2-sided [-29.1 to -7.0]

7. Secondary Outcome: Change From Baseline in Cough Frequency After Cough Challenge Testing in Participants Who Received Gefapixant 100 mg and Placebo (Chronic Cough Participants Only)
Description: An ambulatory cough recording device recorded all sounds chronic cough participants made during cough monitoring to measure the change from baseline in objective cough frequency on the treatment days. A negative change from Baseline was considered to indicate improvement in cough frequency
Time Frame: Baseline and for 24 hours after cough challenge on treatment days
Population: The analyzed population was all treated chronic cough participants who had at least 1 post-dose primary endpoint assessment of cough frequency.
Measure: Least Squares Mean (95% Confidence Interval); unit: Counts/hr
Arm/Group | Gefapixant 100 mg/Chronic Cough | Placebo/Chronic Cough
Number analyzed (Participants) | 24 | 24
Counts/hr | -7.7 [-10.1 to -5.3] | -4.1 [-6.5 to -1.7]
Statistical Analysis 1: Comparison: Gefapixant 100 mg/Chronic Cough vs Placebo/Chronic Cough; Cough Frequency Analysis; Test type: Other; p = 0.0075, Mixed Models Analysis; Mean Difference (Final Values) = -3.6, 95% CI 2-sided [-6.2 to -1.0]

8. Secondary Outcome: Percentage of Participants Who Experienced One or More Adverse Events During Study Treatment and Follow up
Description: A secondary endpoint of the trial was the percentage of participants receiving gefapixant 100 mg and placebo who had at least 1 adverse event (AE) over 4 days of treatment (including washout periods) in addition to 14 days (+3 days) until a post-treatment follow-up visit. An AE is defined as any untoward medical occurrence in a participant administered study drug and which does not necessarily have to have a causal relationship with this treatment. Any worsening of a preexisting condition that is temporally associated with the use of the study drug is also an AE. The percentage of participants in any treatment group with at least 1 AE was assessed.
Time Frame: Up to Day 18
Population: The analyzed population was all randomized participants who took at least 1 dose of study treatment and had assessment of AE occurrence.
Measure: Number; unit: Percentage of participants
Arm/Group | Gefapixant 100 mg/Healthy | Placebo/Healthy | Gefapixant 100 mg/Chronic Cough | Placebo/Chronic Cough
Number analyzed (Participants) | 12 | 12 | 24 | 24
Percentage of participants | 100.0 | 50.0 | 95.8 | 33.3

9. Secondary Outcome: Percentage of Participants Who Discontinued From the Study Due to an Adverse Event
Description: A secondary endpoint of the trial was the percentage of participants receiving gefapixant 100 mg and placebo who discontinued from the study due to an AE. The percentage of participants who discontinued from the study due to an AE was assessed for days 1-4.
Time Frame: Up to Day 4
Population: The analyzed population was all randomized participants who took at least 1 dose of study treatment and had assessment of discontinuation due to an AE.
Measure: Number; unit: Percentage of participants
Arm/Group | Gefapixant 100 mg/Healthy | Placebo/Healthy | Gefapixant 100 mg/Chronic Cough | Placebo/Chronic Cough
Number analyzed (Participants) | 12 | 12 | 24 | 24
Percentage of participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 18
Arm/Group | Gefapixant 100 mg/Healthy | Placebo/Healthy | Gefapixant 100 mg/Chronic Cough | Placebo/Chronic Cough
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 12/12 | 6/12 | 21/24 | 7/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gefapixant 100 mg/Healthy (N=12) | Placebo/Healthy (N=12) | Gefapixant 100 mg/Chronic Cough (N=24) | Placebo/Chronic Cough (N=24)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 0 (0) | 6 (6) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 3 (3) | 0 (0) | 4 (6) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Oral disorder (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (6) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 6 (6) | 1 (1) | 7 (7) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 9 (9) | 1 (1) | 16 (16) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 6 (6) | 2 (2)
Hypogeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The contents of this protocol and any amendments and results obtained during the course of this study will be kept confidential by the Investigator(s), the Investigator's staff, and IRB. No data collected as part of this study will be utilized in any written work, including publications, without the written consent of Sponsor. These obligations shall in no way diminish such obligations as set forth in the Confidentiality Agreement between the Sponsor and the Investigator(s).